CLINICAL TRIAL: NCT00766935
Title: The Equivalency of the Imp SFB7+ (L-Dex U400) With the Imp XCA Device
Status: Completed | Type: Observational
Sponsor: ImpediMed Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: UQSFB7+-01
Record Dates: First submitted 2008-10-02; First posted 2008-10-06 (Estimated); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Lymphedema
Keywords: Lymphedema; Bioimpedance
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1 - lymphoedema group: Females with previously diagnosed unilateral Lymphoedema of the arm, who have had a mastectomy or breast conservation surgery with axillary sampling or dissection, with or without adjuvant therapy.
- 2 - healthy individuals: Healthy females aged between 18-75 years chosen randomly from the population of Queensland, Australia.

SUMMARY:
The purpose of this project is to prove that the Imp™SFB7+ (L-Dex U400) is equivalent to the Imp™ XCA device in assessing Lymphoedema. The Imp™ XCA device is a simple device capable of assessing Lymphoedema of a single arm. The Imp™SFB7+ (L-Dex U400) is a more complex device capable of assessing Lymphoedema in a larger population of Lymphoedema sufferers. The Imp™SFB7+ (L-Dex U400) will be developed to assess patients with Lymphoedema in their arms or their legs. The Imp™ XCA and Imp™ SFB7 are both TGA approved devices. The Imp™ SFB7+ (L-Dex U400) is similar to the Imp™ SFB7 the changes are to the software and user interface.

DETAILED DESCRIPTION:
When Lymphoedema is present, lymph and other fluids build up in the interstitial spaces of the tissues. This results in an overall increase in the total amount of extracellular fluid (ECF) in the limb, causing swelling. This can be documented by measuring the impedance (opposition) to a low frequency current that has been passed into the limb. Low frequency current travels predominantly through the ECF, where the Lymphoedema manifests. As the fluid builds up in the limb, the impedance to the current decreases and it is in this way that low frequency bioimpedance is able to assess Lymphoedema.

Multi-frequency bio-impedance analysis otherwise known as Bioimpedance Spectroscopy (BIS) has been reported to be effective for the measurement of ECF and sub clinical changes in ECF to predict the onset of Lymphoedema in the arms in studies conducted by Cornish et al. It has been reported by Warren et al that BIS can be used as a reliable and accurate tool for documenting presence of lymphoedema in patients with wither upper- or lower-extremity swelling.

The Imp™ XCA device uses an "impedance ratio" methodology to assess unilateral Lymphoedema of the arm. By this method the unaffected arm acts as an internal and subject specific control. The Imp SFB7+ (L-Dex U400) uses the same principles but at a lower frequency. This study is designed to show the equivalence of the 2 devices in assessing unilateral Lymphoedema of the arm.

ELIGIBILITY:
Inclusion Criteria:

Groups 1 and 2

* Be female between the ages of 18-75 years.
* Self-describe general health as satisfactory.
* Understand the proposed study and be willing and fully able to comply with the study procedures.
* Be a willing participant and be capable of giving and has given informed written consent for entry into the study.

Group 1

* Have been previously diagnosed, by current clinical practice, as having unilateral Lymphoedema of the arm of any severity.
* Have had a mastectomy or breast conservation surgery with axillary sampling or dissection, with or without adjuvant therapy.

Exclusion Criteria:

* Have a known heart condition or an implantable device such as a pacemaker or ICD.
* Have a metallic surgical implant (e.g. total hip replacement) not including small implants such as sternal wires or surgical staples.
* Suffer from a renal disorder.
* Be taking diuretic medications.
* Have consumed large amounts of alcohol or caffeinated beverages within six hours of the study.
* Have undertaken excessive exercise within two hours of BIA.
* Have a reported fever of > 38oC at time of screening.
* Be currently in the fourth week of the menstrual cycle.
* Be pregnant or currently breastfeeding.
* Be a relative of any member of study staff or is an employee or a relative of an employee of ImpediMed Ltd.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Group 1 - Primary care clinic Group 2 - Community sample
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2007-11; Primary Completion 2007-12 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Substantial equivalence of the SFB7+ (L-Dex U400) to XCA in the assessment Lymphoedema | Single point measure
  Observation of difference between L-Dex values of lymphoedema population compared to healthy individuals

CONTACTS AND LOCATIONS:
Overall Officials: Robyn Box, PhD, Principal Investigator — Queensland Lymphoedema and Breast Oncology Physiotherapy
Locations (1):
- Queensland Lymphoedema and Breast Oncology Physiotherapy, Brisbane, Queensland, Australia